CLINICAL TRIAL: NCT03399734
Title: A Randomized, Open-Label, Crossover Study to Demonstrate Bioequivalence Between a 4-mg Dose of Fine Granules of Perampanel and a 4-mg Tablet of Perampanel in Healthy Japanese Subjects
Brief Title: Bioequivalence Study Between a 4-mg Dose of Fine Granules of Perampanel and a 4-mg Tablet of Perampanel in Healthy Japanese Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eisai Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: E2007-J081-053
Record Dates: First submitted 2018-01-08; First posted 2018-01-16 (Actual); Last update posted 2018-10-29 (Actual); Status verified 2018-01

CONDITIONS: Healthy Participants
Keywords: Perampanel; Bioequivalence; fine granules; E2007; Japanese
MeSH Terms: interventions — perampanel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment A (Experimental): 4 milligrams (mg) perampanel tablet
  Interventions: Drug: Perampanel
- Treatment B (Experimental): 4 mg perampanel fine granules
  Interventions: Drug: Perampanel

INTERVENTIONS:
Drug: Perampanel — Single oral dose of 1 x 4-mg perampanel tablet
  Other Names: E2007
  Arms: Treatment A
Drug: Perampanel — Single 4-mg dose of perampanel fine granules
  Other Names: E2007
  Arms: Treatment B

SUMMARY:
This study will be conducted to demonstrate the bioequivalence between a single 4 milligram (mg) dose of fine granules of perampanel and a single 4 mg tablet of perampanel.

ELIGIBILITY:
Inclusion Criteria

Participants must meet all of the following criteria to be included in this study:

* Non-smoking, male or female age ≥20 years and ≤45 years old at the time of obtaining written informed consent. To be considered non-smokers, participants must have discontinued smoking from Screening before first dosing.
* Body Mass Index ≥18.5 and <25.0 kilograms per meters squared at Screening

Exclusion Criteria

Participants who meet any of the following criteria will be excluded from this study:

* Females who are breastfeeding or pregnant at Screening or Baseline
* Clinically significant illness that requires medical treatment within 8 weeks or a clinically significant infection that requires medical treatment within 4 weeks before first dosing
* Evidence of disease that may influence the outcome of the study within 4 weeks before first dosing
* Any history of gastrointestinal surgery that may affect pharmacokinetic profiles of perampanel at Screening
* Any clinically abnormal symptom or organ impairment found by medical history at Screening, and physical examinations, vital signs, electrocardiogram (ECG) finding, or laboratory test results that require medical treatment at Screening
* A prolonged QT/QT corrected interval (QT interval, Fridericia correction >450 milliseconds) as demonstrated by a repeated ECG at Screening or Baseline

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2017-12-18 (Actual); Primary Completion 2018-03-09 (Actual); Study Completion 2018-03-09 (Actual)

PRIMARY OUTCOMES:
Maximum observed concentration (Cmax) | 0-168 hours postdose of Treatment Period 1 and Treatment Period 2
Area under the concentration-time curve from zero time to 168 hours (AUC[0-168h]) | 0-168 hours postdose of Treatment Period 1 and Treatment Period 2

SECONDARY OUTCOMES:
Time at which the highest drug concentration occurs (tmax) | 0-168 hours postdose of Treatment Period 1 and Treatment Period 2
Lag time (tlag) | 0-168 hours postdose of Treatment Period 1 and Treatment Period 2
  tlag is the time delay between drug administration and the onset of drug absorption.
Area under the concentration-time curve from zero time to 72 hours (AUC[0-72h]) | 0-72 hours postdose of Treatment Period 1 and Treatment Period 2
Area under the concentration-time curve from zero time to time of the last quantifiable concentration (AUC[0-t]) | 0-168 hours postdose of Treatment Period 1 and Treatment Period 2
Area under the concentration-time curve from zero time extrapolated to infinite time (AUC[0-inf]) | 0-168 hours postdose of Treatment Period 1 and Treatment Period 2
Terminal phase rate constant (λz) | 0-168 hours postdose of Treatment Period 1 and Treatment Period 2
Terminal elimination phase half-life (t1/2) | 0-168 hours postdose of Treatment Period 1 and Treatment Period 2
Mean residence time (MRT) | 0-168 hours postdose of Treatment Period 1 and Treatment Period 2

CONTACTS AND LOCATIONS:
Locations (1):
- Eisai Trial Site, Toshima-ku, Tokyo, Japan